CLINICAL TRIAL: NCT04102930
Title: UK GCA Consortium: Clinical and Immunogenetic Characterization of Giant Cell Arteritis (GCA) and Polymyalgia Rheumatica (PMR)
Brief Title: Clinical and Immunogenetic Characterization of Giant Cell Arteritis (GCA) and Polymyalgia Rheumatica (PMR)
Status: Recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Ann Morgan, Professor of Molecular Rheumatology and Honorary Consultant Rheumatologist, University of Leeds
Other Study IDs: MM05/7037
Record Dates: First submitted 2019-07-30; First posted 2019-09-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Giant Cell Arteritis; Polymyalgia Rheumatica
MeSH Terms: conditions — Giant Cell Arteritis; Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Serum, plasma, cellular and subcellular fractions of blood, urine or arterial tissue, DNA, RNA, proteins and metabolites
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective: A patient who has a diagnosis of GCA or PMR
- Prospective: Patient with suspected GCA and PMR

SUMMARY:
A multi-centre observational study recruiting prospective and retrospective cohorts of patients with polymyalgia rheumatica (PMR) and giant cell arteritis (GCA). The primary aim is to find genetic determinants of GCA and PMR susceptibility, in order to yield novel insights into disease pathogenesis. A subset of the retrospective cohort is also enrolled in a post-marketing surveillance registry of patients eligible for, or receiving tocilizumab, to treat their relapsing or refractory GCA.

DETAILED DESCRIPTION:
Giant cell arteritis (GCA), also known as temporal arteritis, is the most common form of primary systemic vasculitis, with up to 75,000 cases a year identified in the EU and US. It occurs almost exclusively in people over the age of 50 years and is considered to be a medical emergency. If not treated with high-dose glucocorticoids immediately, the thickening of the inflamed blood vessel wall can cause irreversible visual loss or stroke. GCA can lead to significant morbidity across a variety of systems, due to both the disease, and complications of treatment. Diagnosis may be confirmed with a temporal artery biopsy, imaging (e.g. USS/CT/MRA/PET-CR) or based on clinical signs (e.g. erythrocyte sedimentation rate) and symptoms (e.g. a new headache, jaw claudication, visual disturbances, temporal artery abnormality such as tenderness or decreased pulsation) .

Polymyalgia rheumatica (PMR) is characterised by inflammatory limb-girdle pain with early morning stiffness, and a systemic inflammatory response demonstrated by elevated inflammatory markers.

The UK GCA Consortium is a multi-centre observational study, the main arms of which recruit prospective (participants with suspected GCA) and retrospective cohorts (participants with confirmed GCA diagnosis). Analysis of data collected on these cohorts will help achieve the primary aim of finding genetic determinants of GCA and PMR susceptibility, in order to yield novel insights into disease pathogenesis. Secondary aims, and their associated analyses, are as follows:

* Phenotype: characterising GCA and PMR subtypes, based on clinical features; imaging; cells; subcellular fractions and molecules in the circulation and/or arterial tissue; genetic/epigenetic/transcriptomic/proteomic or metabolomics factors, including next generation sequencing (whole exome sequencing) of selected cases.
* Life impact: determining what aspects of the disease and treatments affect patients' quality of life, as assessed by patient-reported outcomes.
* Long-term outcomes: characterising prognosis of GCA and PMR - both effects of the disease and its treatment - by longitudinal follow-up through electronic linkage to health records.
* Exploratory analyses: exploring the potential role of environmental factors and co-morbidities on phenotype and outcomes.
* Diagnosis, prognosis: improving diagnosis of GCA and PMR, and identifying factors that predict diagnosis, such as diagnostic clinical features, and prognostic and diagnostic biomarkers.
* Disease activity: monitoring participants who commence a synthetic or biological disease-modifying anti-rheumatic drug (s/bDMARD). Finding a biomarker for GCA and PMR disease activity, which might be clinically useful in helping to optimise steroid and s/bDMARD treatments for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing to self-identify an ethnic group, such as Caucasian, Asian, Afro-Caribbean.
* Have a firm clinical diagnosis of GCA or PMR, or (for patients identified prospectively) GCA or PMR should be more likely than any alternative explanation for the patient's symptoms.
* Able and willing to give informed consent. Patients will be 50 years of age or over, unless both biopsy-proven and a clinically classical case of GCA.

Exclusion Criteria:

• Patient unwilling or unable to give fully informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients predominantly recruited from secondary but can be identified and/or recruited in primary care.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2005-06-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome for genetic susceptibility studies: | At baseline
  Diagnosis of GCA (or PMR), confirmed by a specialist (e.g. rheumatologist, ophthalmologist) with relevant expertise.

SECONDARY OUTCOMES:
Phenotype | At baseline
  Clinical phenotype or subtype of GCA/PMR based on disease features and imaging undertaken as part of routine clinical practice, and on research tests, such as imaging performed for research purposes, cells, subcellular fractions and molecules in the circulation and/or arterial tissue and genetic/ epigenetic/ transcriptomic/ proteomic or metabolomic factors, including next generation sequencing (whole exome sequencing) of selected cases.
Life impact questionnaires | At baseline
  Assessment of the impact the disease and treatment has on the patients' lives as reported by the patient
Long term outcomes | At baseline
  Longitudinal follow-up of patients (as far as is possible from medical and electronic records and without requiring additional study visits) to define prognosis/disease outcomes, such as ischaemic manifestations, aneurysm formation, duration of steroid therapy, disease flares, complications related to steroid therapy.
Diagnosis of GCA/PMR | Through study completion, an average of 1 year
  Diagnosis in patients presenting with suspected GCA/PMR (prospective study).
Exploratory analyses | At baseline
  To investigate role of genetics, environmental factors (e.g. diet and sunlight) and co-morbidities (e.g. periodontal disease) on disease phenotype and outcome as assessed by the patient-administered questionnaires.
Disease activity defined as an increase in clinical and patient reported activity of disease | At baseline
  Participants commencing a synthetic or biological disease modifying anti-rheumatic drug with or without additional steroid therapy will have their disease activity assessed.
Proteomic and genomic analyses on serum, plasma and urine samples. | At baseline
  A variety of 'omic technologies will be applied to cell populations isolated from the blood and/or routine diagnostic arterial biopsies, including, but not limited to, RNASeq and a variety of proteomic approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Morgan, Principal Investigator — University of Leeds
Locations (76):
- United Kingdom (76):
  - Queen Elizabeth The Queen Mother Hospital, Canterbury, Kent
  - Whiston Hospital, Prescot, Merseyside
  - Nevill Hall Hospital, Aneurin Bevan University Health Board, Abergavenny
  - Stoke Mandeville Hospital, Buckinghamshire Healthcare NHS Trust, Aylesbury
  - Betsi Cadwaladr University Health Board, Bangor
  - Barnsley Hospital, Barnsley Hospital NHS Foundation Trust, Barnsley
  - Basildon University Hospital, Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon
  - Basingstoke and North Hampshire Hospital, Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Royal National Hospital for Rheumatic Diseases, Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Birmingham Heartlands Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Bristol Royal Infirmary, University Hospitals Bristol NHS Foundation Trust, Bristol
  - Queen's Hospital, University Hospitals of Derby and Burton NHS Foundation Trust, Burton-on-Trent
  - West Suffolk Hospital, West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Addenbrookes Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Chelsea and Westminster Hospital, Chelsea and Westminster Hospital NHS Foundation Trust, Chelsea
  - West Middlesex University Hospital, Chelsea and Westminster Hospital NHS Foundation Trust, Chelsea
  - Ashford and St Peter's Hospitals, Ashford & St Peter's Hospitals NHS Foundation Trust, Chertsey
  - Countess of Chester Hospital, Countess of Chester NHS Foundation Trust, Chester
  - Christchurch Hospital, University Hospitals Dorset NHS Foundation Trust, Christchurch
  - Croydon University Hospital, Croydon Health Service NHS Trust, Croydon
  - Darlington Memorial Hospital, County Durham and Darlington NHS Foundation Trust, Darlington
  - Royal Derby Hospital, University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - Doncaster Royal Infirmary, Doncaster and Bassetlaw Hospitals NHS Foundation Trust, Doncaster
  - Ninewells Hospital and Medical School, NHS Tayside, Dundee
  - Royal Devon and Exeter Hospital, Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Frimley Park Hospital, Frimley Park Hospital NHS Foundation Trust, Frimley
  - Gateshead Queen Elizabeth Hospital, Gateshead Health NHS Foundation Trust, Gateshead
  - Inverclyde Royal Hospital, NHS Greater Glasgow and Clyde, Glasgow
  - Royal Alexandra Hospital, NHS Greater Glasgow and Clyde, Glasgow
  - Vale of Leven Hospital, NHS Greater Glasgow and Clyde, Glasgow
  - James Paget Hospital, James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Royal Surrey County Hospital, Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Harrogate and District Hospital, Harrogate and District NHS Foundation Trust, Harrogate
  - Hull Royal Infirmary, Hull and East Yorkshire NHS Trust, Hull
  - Ipswich Hospital, East Suffolk and North Essex NHS Foundation Trust, Ipswich
  - Airedale General Hospital, Airedale NHS Foundation Trust, Keighley
  - Westmorland General Hospital, University Hospitals of Morecambe Bay NHS Foundation Trust, Kendal
  - The Queen Elizabeth Hospital, The Queen Elizabeth Hospital Kings Lynn NHS Foundation Trust, Kings Lynn
  - Royal Lancaster Infirmary, University Hospitals of Morecambe NHS Foundation Trust, Lancaster
  - Chapel Allerton Hospital, Leeds Teaching Hospitals NHS Foundation Trust, Leeds
  - Leicester Royal Infirmary, University Hospitals of Leicester NHS Trust, Leicester
  - Aintree University Hospital, Aintree University Hospitals NHS Trust, Liverpool
  - Royal Glamorgan Hospital, Cwm Taf University Health Board, Llantrisant
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - King's College Hospital, King's College Hospital NHS Foundation Trust, London, London
  - Royal Free Hospital, Royal Free NHS Foundation Trust, London
  - St George's Hospital, St George's University Hospitals NHS Foundation Trust, London
  - University College London Hospital, University College London NHS Foundation Trust, London
  - Manchester Royal Infirmary, Manchester University NHS Foundation Trust, Manchester
  - Arrowe Park Hospital, Wirral University Hospital NHS Foundation Trust, Metropolitan Borough of Wirral
  - Freeman Hospital, The Newcastle-upon-Tyne Hospitals NHS Foundation Trust, Newcastle
  - North Tyneside General Hospital, Northumbria Healthcare NHS Foundation Trust, North Shields
  - Northampton General Hospital, Northampton General Hospital NHS Trust, Northampton
  - Norfolk and Norwich University Hospital, Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Queens Medical Centre, Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford Nuffield Orthopaedic Centre, Oxford University Hospitals NHS Trust, Oxford
  - Peterborough City Hospital, North West Anglia NHS Foundation Trust, Peterborough
  - Derriford Hospital, University Hospital Plymouth NHS Trust, Plymouth
  - Poole Hospital, University Hospitals Dorset NHS Foundation Trust, Poole
  - Minerva Health Centre, Lancashire and South Cumbria NHS Foundation Trust, Preston
  - Royal Preston Hospital, Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Salford Royal Hospital, Salford Royal NHS Foundation Trust, Salford
  - Scarborough General Hospital, York and Scarborough Teaching Hospitals NHS Foundation Trust, Scarborough
  - Southend University Hospital, Southend University Hospital NHS Foundation Trust, Southend-on-Sea
  - Lister Hospital, East and North Hertfordshire NHS Trust, Stevenage
  - Haywood Hospital, Midlands Partnership NHS Foundation Trust, Stoke-on-Trent
  - Great Western Hospital, The Great Western Hospitals NHS Foundation Trust, Swindon
  - Torbay Hospital, Torbay and South Devon NHS Foundation Trust, Torquay
  - Royal Cornwall Hospital, Royal Cornwall Hospitals NHS Trust, Truro
  - Pinderfields Hospital, Mid Yorkshire Hospitals NHS Trust, Wakefield
  - Warrington Hospital, Warrington and Halton Hospitals NHS Foundation Trust, Warrington
  - Warwick Hospital, South Warwickshire NHS Foundation Trust, Warwick
  - Royal Hampshire County Hospital, Hampshire Hospitals NHS Foundation Trust, Winchester
  - University Hospital Wishaw, NHS Lanarkshire, Wishaw
  - York Hospital, York and Scarborough Teaching Hospitals NHS Foundation Trust, York